CLINICAL TRIAL: NCT05431673
Title: Efficacy Of Doxycycline & Versus Rifampin In Treatment Of Rhinoscleroma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdullah Mohamad Omar, Resident of otorhinolaryngology department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Doxycycline in Rhinoscleroma
Record Dates: First submitted 2021-12-14; First posted 2022-06-24 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Rhinoscleroma
Keywords: doxycycline
MeSH Terms: conditions — Rhinoscleroma | interventions — Doxycycline; Ciprofloxacin; Rifampin

STUDY DESIGN:
Intervention Model Description: 3 Groups A will receive Doxycycline B will receive Ciprofloxacin and Doxycycline C will receive Rifampin
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Doxycycline (Active Comparator): • Subjects in this group will be treated with Doxycycline (100mg/day for 8 weeks).[1]
  Interventions: Drug: Doxycycline
- Doxycycline & Ciprofloxacin (Active Comparator): • Subjects in this group will be treated with combination of Doxycycline (100mg/day for 8 weeks) & Ciprofloxacin (250mg twice daily for 4 weeks).[1]
  Interventions: Drug: Doxycycline; Drug: Ciprofloxacin
- Rifampicin (Active Comparator): • Subjects in this group will be treated with Rifampicin (600mg/day for 6 weeks)
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 100mg/day for 6 weeks used as single or combination treatment for Rhinoscleroma
  Arms: Doxycycline; Doxycycline & Ciprofloxacin
Drug: Ciprofloxacin — Ciprofloxacin 500mg/day for 4 weeks used as single or combination treatment for Rhinoscleroma
  Arms: Doxycycline & Ciprofloxacin
Drug: Rifampin — Rifampin 600mg/day for 6 weeks used as single or combination treatment for Rhinoscleroma
  Arms: Rifampicin

SUMMARY:
The study is conducted To evaluate the Efficacy of Doxycycline (alone and in combination with Ciprofloxacin) as an alternative to the regular regimen in treating rhinoscleroma, especially for cases with contraindication to the use of one or more of the regularly used drugs.

DETAILED DESCRIPTION:
Rhinoscleroma is a chronic granulomatous disease endemic in many eastern countries including Egypt, Its causative agent is a gram-negative bacillus, Klebsiella rhinoscleromatis. Low socioeconomic populations are the most affected.. There are four known stages of the lesion. The first of which the 'Catarrhal stage' with purulent rhinorrhea, then there is the 'Atrophic stage' with a picture similar to that of atrophic rhinitis. The next is the 'Hypertrophic' or 'Granulomatous' stage where there are bluish red rubbery nodules in any part along the distribution of the disease, and eventually the 'Fibrotic' or 'Sclerotic' stage with stenosis deformity and loss of functions of the parts affected. Examples of commonly used drugs are 'Rifampicin' which is the most commonly used drug exhibits good results but the need for close monitoring for fear of toxicity is the only limitation to its use, Ciprofloxacin' is another Antibiotic with special efficacy as it has good tissue penetration & produces high concentrations in respiratory tract secretions. Recently 'Doxycycline' has been approved to be used in rhinoscleroma which has the advantage of not only easier dosing but also better patient compliance as it's used for a shorter course (6 weeks) compared to most other drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included after confirmation by histopathological examination.
* Patients presented in active stages of the disease.
* Patients between 18-70 years.

Exclusion Criteria:

* Any granulomatous lesion or features suggestive of rhinoscleroma associated with any other nasal lesions like syphilis, leprosy and tuberculosis were excluded.
* Patients below 18 years and above 70 years.
* Biopsy-negative cases.
* Patients in Atrophic or Sclerotic Stages of the disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-08-21 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients showing post treatment histopathologic resolution | 8 months from the start of treatment
  Comparing Histopathologic changes pre and post intervention for the 3 groups and the number of participants whose post treatment biopsy show histopathologic resolution will be measued as percentage to the total number of participants in each group

SECONDARY OUTCOMES:
Nasal Symptoms | 8 months from the start of treatment
  All participants will be asked to score 5 nasal symptoms (nasal congestion/obstruction, anterior rhinorrhea, posterior rhinorrhea, loss of smell and facial pain.) from 0 to 4.
  0= no symptoms
  1. mild symptoms
  2. moderate symptoms
  3. sever symptoms
  4. very sever symptoms this score will be assessed at the screening visit & follow up visits at 8 weeks , 6 months.
  the total five-symptom score obtained will be the sum of the individual symptoms(0-20)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed AbdelAleem, PhD, Study Director — Assiut University

REFERENCES:
- [Background] Kallapa S, Sarkar SR, Shankar MG. Effectiveness of ciprofloxacin vs. doxycycline in treatment of rhinoscleroma- A case-control study. J. Evid. Based Med. Healthc. 2017; 4(20), 1165-1168
- [Background] Abou-Seif SG, Baky FA, el-Ebrashy F, Gaafar HA. Scleroma of the upper respiratory passages: a CT study. J Laryngol Otol. 1991 Mar;105(3):198-202. doi: 10.1017/s0022215100115348. PMID 2019806
- [Background] Badia L, Lund VJ. A case of rhinoscleroma treated with ciprofloxacin. J Laryngol Otol. 2001 Mar;115(3):220-2. doi: 10.1258/0022215011907028. PMID 11244532
- [Background] Cone LA, Barton SM, Woodard DR. Treatment of scleroma with ceforanide. Arch Otolaryngol Head Neck Surg. 1987 Apr;113(4):374-6. doi: 10.1001/archotol.1987.01860040036012. PMID 3814386
- [Background] Jage M, Rambhia KD, Khopkar US. Efficacy of doxycyclin monotherapy in treating rhinoscleroma. Indian J Drugs Dermatol 2018;4:23-5
- [Background] Menzies D, Benedetti A, Paydar A, Martin I, Royce S, Pai M, Vernon A, Lienhardt C, Burman W. Effect of duration and intermittency of rifampin on tuberculosis treatment outcomes: a systematic review and meta-analysis. PLoS Med. 2009 Sep;6(9):e1000146. doi: 10.1371/journal.pmed.1000146. Epub 2009 Sep 15. PMID 19753109